CLINICAL TRIAL: NCT03193554
Title: Diagnostic Value of microRNA 210 In Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yousra M Farghaly, principal investigator, Assiut University
Other Study IDs: D V O MicroRNA210 I PET
Record Dates: First submitted 2017-06-18; First posted 2017-06-21 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pre-eclampsia is a disorder of pregnancy characterized by hypertension (defined as systolic blood pressure 140mmHg or diastolic blood pressure ⩾90 mmHg) and proteinuria (300 mg or greater in a 24 h urine specimen and/or protein to creatinine ratio of > 0.30) . The disorder usually occurs after 20 weeks of pregnancy and worsens over time. Risk factors for pre-eclampsia include: obesity, prior hypertension, older age, and diabetes mellitus, primigravida and pregnant women with multiple gestation .

Healthy women pregnancy can be associated with resistance to the action of insulin on glucose uptake and utilization. Insulin Resistance (IR) is defined as decreased ability of target tissues such as liver, adipose tissue and muscle to respond to normal circulating concentrations of insulin. Insulin Resistance can be a result of a number of factors such as defective molecular structure of insulin, defective receptor functioning or defective signal transduction pathway .

Preeclampsia is associated with increased expression of Tumor necrosis Factor α and other inflammatory marker which causes Insulin Resistance. Increased Insulin Resistance leads to dyslipidemia that can worsen the placental ischemia leading to vicious cycle of ischemia-inflammation-Insulin Resistance-dyslipidemia-ischemia . Insulin resistance has also been hypothesized to contribute to the pathophysiology of preeclampsia. Compared to women who have normotensive pregnancies, women who develop preeclampsia are more insulin resistant prior to pregnancy .

The recognition that specific miRNAs are induced by hypoxia and are commonly dysregulated in preeclampsia raises the possibility that such miRNAs mediate the adverse effects of placental hypoxia in preeclampsia. MiRNAs present in maternal blood may have the potential to be used as biomarkers, as they are relatively stable and tissue specific . It was found that mir-210 is induced in patients with pre-eclampsia, whether mir-210 contributes to the pathogenesis of pre-eclampsia, a complex disorder widely believed to be associated with placental hypoxia .

DETAILED DESCRIPTION:
Pre-eclampsia is a disorder of pregnancy characterized by hypertension (defined as systolic blood pressure ⩾140 mmHg or diastolic blood pressure ⩾90 mmHg) and proteinuria (300 mg or greater in a 24 h urine specimen and/or protein to creatinine ratio of > 0.30) . The disorder usually occurs after 20 weeks of pregnancy and worsens over time . Preeclampsia is routinely screened during prenatal care .

In severe disease there may be red blood cell breakdown, a low blood platelet count, impaired liver function, kidney dysfunction, swelling, shortness of breath due to fluid in the lungs, or visual disturbances. Pre-eclampsia increases the risk of poor outcomes for both the mother and the baby . If left untreated, it may result in seizures at which point it is known as eclampsia or HELLP syndrome (hemolysis ,elevated liver enzymes , low platelets ) .

The clinical features of preeclampsia are caused by systemic maternal endothelial dysfunction resulting from a combination of preexisting maternal risk factors and abnormal placental development. Risk factors for pre-eclampsia include: obesity, prior hypertension, older age, and diabetes mellitus . It is also more frequent in a woman's first pregnancy and if she is carrying twins. The underlying mechanism involves abnormal formation of blood vessels in the placenta amongst other factors .

These maternal characteristics may contribute to oxidative stress, inflammation and vascular dysfunction, all of which have been implicated in the etiology of preeclampsia .

Healthy women pregnancy can be associated with resistance to the action of insulin on glucose uptake and utilization . Insulin Resistance is defined as decreased ability of target tissues such as liver, adipose tissue and muscle to respond to normal circulating concentrations of insulin. Insulin Resistance can be a result of a number of factors such as defective molecular structure of insulin, defective receptor functioning or defective signal transduction pathway .

Many maternal hormones and factors play role in causation of Insulin Resistance during pregnancy such as increased levels of serum cortisol, Tumor necrosis factor α , can interrupt the insulin signaling pathway and can lead to Insulin Resistance during normal pregnancy .

Women with increased Insulin Resistance are more prone to develop preeclampsia and gestational diabetes. Preeclampsia is associated with increased expression of Tumor necrosis factor α and other inflammatory marker which causes Insulin Resistance. Increased Insulin Resistance leads to dyslipidemia that can worsen the placental ischemia leading to vicious cycle of ischemia-inflammation-Insulin Resistance-dyslipidemia-ischemia .

Insulin resistance has also been hypothesized to contribute to the pathophysiology of preeclampsia. Compared to women who have normotensive pregnancies, women who develop preeclampsia are more insulin resistant prior to pregnancy .

Early reliable markers for preeclampsia development is the involvement of microRNA in the pathogenesis and its possible role as an early biomarker for disease development. MicroRNAs (miRNAs) are a series of small (18-24 nt) endogenous noncoding single-stranded RNAs, which can regulate gene expression post transcriptionally by a nonperfect pairing of 6-8 nucleotides with target mRNAs . It is currently estimated that up to 30% of human genes may contain miRNAs' binding sites, which suggested a potential role of microRNAs as central regulators in the control of gene expression .

MicroRNAs have been implicated in a variety of human diseases, such as cardiovascular disease, primary muscular disorders, and cancer. In addition, miRNAs have been reported involved in regulating pregnancy process .

The human placenta exhibits a specific microRNA expression pattern that dynamically changes during pregnancy and is reflected in the maternal plasma .

The recognition that specific microRNAs are induced by hypoxia and are commonly dysregulated in preeclampsia raises the intriguing possibility that such microRNAs mediate the adverse effects of placental hypoxia in preeclampsia. The connection between microRNAs, adipose tissue, and insulin resistance may have a role in gestational diabetes mellitus pathophysiology. microRNAs present in maternal blood may have the potential to be used as biomarkers, as they are relatively stable and tissue specific .

MicroRNA 210 is identified as a unique hypoxia induced miRNA that is universally induced in various cell types. Using microRNA microarray it was found that microRNA 210 is overexpressed in placental tissue derived from patients with pre-eclampsia .

It was found whether microRNA 210 contributes to the pathogenesis of pre-eclampsia, a complex disorder widely believed to be associated with placental hypoxia. The results show that microRNA 210 is induced in patients with pre-eclampsia and in hypoxia treated trophoblast cells .

It has been found that microRNA 210 levels are dramatically increased in the placental tissue derived from patients with preeclampsia. In this issue, MicroRNA 210 levels in plasma from preeclampsia patients were significantly higher than those in gestational healthy controls. Furthermore, the expression levels of microRNA 210 seemed to correlate well with disease severity, suggesting a potential role of circulating microRNA 210 as novel biomarker for the diagnosis of preeclampsia.

ELIGIBILITY:
Inclusion Criteria :Pregnant females that admitted to Women's Health Hospital and they will be divided as follow:

* Group 1: Pregnant women with insulin resistance .
* Group 2: Healthy pregnant women as control group .

Exclusion Criteria:

- 1- Female patients with any other type of malignant or benign tumours should be excluded from our study.

2- Past history of chemotherapy or surgical treatment of cancer. 3-Women who diagnosed as preeclamptic or diabetic

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Study Population: Pregnant women in second trimster divided into 2 groups :
  1. Physiological high risk factor for preeclampsia .
  2. Pregnant women with high insulin resistance.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of MicroRNA 210 in preeclampsia | 1 Year

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - ASSIUT University, Asyut
  - Assiut Unversity, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Jameil N, Aziz Khan F, Fareed Khan M, Tabassum H. A brief overview of preeclampsia. J Clin Med Res. 2014 Feb;6(1):1-7. doi: 10.4021/jocmr1682w. Epub 2013 Dec 13. PMID 24400024
- [Background] Bueno MJ, Perez de Castro I, Malumbres M. Control of cell proliferation pathways by microRNAs. Cell Cycle. 2008 Oct;7(20):3143-8. doi: 10.4161/cc.7.20.6833. Epub 2008 Oct 20. PMID 18843198
- [Background] Eiland E, Nzerue C, Faulkner M. Preeclampsia 2012. J Pregnancy. 2012;2012:586578. doi: 10.1155/2012/586578. Epub 2012 Jul 11. PMID 22848831
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Morales Prieto DM, Markert UR. MicroRNAs in pregnancy. J Reprod Immunol. 2011 Mar;88(2):106-11. doi: 10.1016/j.jri.2011.01.004. Epub 2011 Feb 25. PMID 21353310
- [Background] Roberts JM, Lain KY. Recent Insights into the pathogenesis of pre-eclampsia. Placenta. 2002 May;23(5):359-72. doi: 10.1053/plac.2002.0819. PMID 12061851
- [Background] Steegers EA, von Dadelszen P, Duvekot JJ, Pijnenborg R. Pre-eclampsia. Lancet. 2010 Aug 21;376(9741):631-44. doi: 10.1016/S0140-6736(10)60279-6. Epub 2010 Jul 2. PMID 20598363